CLINICAL TRIAL: NCT02452541
Title: Early Determination of Neurological Prognosis in ICU Patients With Severe Traumatic Brain Injury: The TBI-Prognosis Multicenter Prospective Study
Brief Title: TBI-Prognosis Multicenter Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government); Canadian Critical Care Trials Group (Other)
Responsible Party: Principal Investigator, Alexis Turgeon, MD MSc FRCPC, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PEJ-679
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Critically ill Patients; Death; Head Injury; TBI-Prognosis; Critical Care Medicine; Withdrawal of Life Sustaining Therapy; Prognosis; Prognostic Evaluation; Outcome Research; Mortality; Decision-making
MeSH Terms: conditions — Brain Injuries, Traumatic; Death; Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prognostic evaluation (Other): Prognostic tests/exams performed according to a determined schedule during the acute phase of care following admission in the intensive care unit.
  Interventions: Other: Prognostic tests

INTERVENTIONS:
Other: Prognostic tests — * Brain CT-Scan on day 1, 3 and 7
  * Brain MRI on day 7
  * SomatoSensory Evoked Potentials on day 7
  * Electroencephalogram on day 7
  * Serum biomarkers on day 1, 3 and 7
  * Daily clinical exams

SUMMARY:
Severe traumatic brain injury (TBI) is the leading cause of death and disability among people under 45 years of age and a major public health problem. Although management of severe TBI patients has gradually improved with the establishment of intensive care units (ICU) and the development of practice guidelines, mortality is still high - ranging from 30 to 50% - with 30% of survivors suffering from severe neurological sequelae such as neurovegetative states. Families and medical teams are frequently called upon to determine reasonable and appropriate goals of care for brain injured patients. They may have to consider high intensity of care, but also the withdrawal of life-sustaining therapies in accordance with patient wishes. Physicians involved in the care of severe traumatic brain injury have expressed serious concerns about hasty decisions made in the absence of appropriate evidence of unfavourable prognosis. The purpose of the TBI-Prognosis study is to develop a prognostic model by using a multimodal approach of different prognostic indicators and their evolution over time in the acute phase of care. The results of this study will provide better objective information that will facilitate the shared-decision making-process with families and relatives.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) with severe blunt TBI admitted to the ICU
* All patients with a GCS ≤ 8 after initial resuscitation

Exclusion Criteria:

* Anticipated being on mechanical ventilation for < 48 hour period due to an altered level of consciousness related to the TBI plus another potentially reversible factor (i.e. drugs, substance abuse, excessive sedation, etc.).
* Solid malignancy with a life expectation <12 months
* Liver cirrhosis Child C
* Chronic heart failure (NYHA class IV)
* End-stage chronic respiratory disease (O2 dependent)
* End-stage renal disease (initiated or expectant chronic dialysis or to be expected)
* Previous neurologic disorder with abnormal findings (such as a mass lesion) on radiological imaging (CT-scan, MRI) or electrophysiological tests (EEG, SSEP) (such as previous uncontrolled epilepsy, significant stroke, previous or acute concomitant spinal cord injury, etc)
* Patients with no fixed address will be excluded because of the difficult follow-up
* Physician refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2013-04; Primary Completion 2017-02 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended | 12 months

SECONDARY OUTCOMES:
EuroQuol - EQ-5D-5L | 12 months
Glasgow Outcome Scale Extended | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Turgeon, MD MSc FRCPC, Principal Investigator — CHU de Quebec Research Center
Locations (17):
- Canada (17):
  - Foothills Health Sciences Centre, Calgary, Alberta
  - Capital Health - Royal Alexandra Hospital, Edmonton, Alberta
  - Capital Health - University Of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Winnipeg Health Sciences Center, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - ST. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - CHU de Québec - Hôpital de l'Enfant-Jésus, Québec, Quebec
  - CHU Sherbrooke - Hôpital Fleurimont, Sherbrooke, Quebec